CLINICAL TRIAL: NCT01281514
Title: Phase I Study of Carboplatin, Pegylated Liposomal Doxorubicin (PLD) and Everolimus in Patients With Platinum-Sensitive Epithelial Ovarian, Fallopian Tube or Primary Peritoneal Cancer in First Relapse
Brief Title: A Study of Carboplatin, PLD and Everolimus in Certain Gynecologic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB 10-019; NCI-2011-00055 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); GYN-067 (Other: Fox Chase Cancer Center)
Record Dates: First submitted 2011-01-12; First posted 2011-01-24 (Estimated); Last update posted 2019-07-11 (Actual); Status verified 2019-07

CONDITIONS: Fallopian Tube Cancer; Peritoneal Cavity Cancer; Recurrent Ovarian Epithelial Cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Everolimus; Carboplatin; liposomal doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): See Detailed Description
  Interventions: Drug: everolimus; Drug: carboplatin; Drug: pegylated liposomal doxorubicin hydrochloride; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: everolimus — Given PO
  Other Names: 42-O-(2-hydroxy)ethyl rapamycin; Afinitor; RAD001
Drug: carboplatin — Given IV
  Other Names: Carboplat; CBDCA; JM-8; Paraplat; Paraplatin
Drug: pegylated liposomal doxorubicin hydrochloride — Given IV
  Other Names: CAELYX; Dox-SL; DOXIL; doxorubicin hydrochloride liposome; LipoDox
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as carboplatin and pegylated liposomal doxorubicin hydrochloride (PLD) work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Everolimus may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving carboplatin and PLD together with everolimus may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of everolimus when given together with carboplatin and PLD in treating patients with relapsed ovarian epithelial, fallopian tube, or peritoneal cavity cancer

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximum tolerated dose (MTD) of RAD001 (everolimus) in combination with carboplatin and PLD.

SECONDARY OBJECTIVES:

I. Determine safety/tolerability of the three drug combination of carboplatin, PLD and RAD001 (everolimus).

II. Determine preliminary analysis of anti-tumor activity of this regimen in patients with recurrent ovarian, fallopian tube or primary peritoneal cancers.

OUTLINE: This is a dose-escalation study of everolimus.

Patients receive carboplatin intravenously (IV) and PLD IV on day 1 and everolimus orally (PO) once daily on days 1-28. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 2 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed epithelial ovarian, fallopian tube, or primary peritoneal carcinoma
* Patients must have had exactly one prior platinum/taxane-based chemotherapeutic regimen for management of primary disease, and must be in first relapse; first relapse must occur >= six months from completion of front-line platinum-based therapy; (time measured from last platinum dose; for example, patients receiving a biologic or chemotherapeutic agent after completion of platinum-based therapy as part of upfront therapy would be eligible based on time from last dose of platinum chemotherapy; in this situation, patients must be at least four weeks from last dose of a biologic agent); relapse cannot be based on rising cancer antigen (CA)- 125 alone; there must be radiographic evidence of recurrent disease
* Measurable disease as per Response Evaluation Criteria In Solid Tumors (RECIST) v1.1 criteria or non-measurable disease with symptomatic malignant pleural effusion or malignant ascites; if only site of disease is a pleural effusion, cytologic confirmation of recurrence should be obtained
* Patients must not have any major surgery or radiation therapy within 14 days of start of study treatment
* All acute toxicities from prior therapy with the exception of alopecia must have resolved to =< grade 1
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Absolute neutrophil count (ANC) >= 1500
* Platelets >= 100K
* Serum total bilirubin =< 1.5x upper limit of normal (ULN)
* Serum transaminase (aspartate aminotransferase [AST]/serum glutamic oxaloacetic transaminase [SGOT], alanine aminotransferase [ALT]/serum glutamic pyruvic transaminase [SGPT]) activity =< 2.5 x ULN
* International normalized ratio (INR) =< 1.5 and partial thromboplastin time (PTT) =< 1.5 x ULN for patients who are not being treated with therapeutic anticoagulation; therapeutic or prophylactic anticoagulation is allowed if a patient has been on a stable dose of low molecular weight (LMW) heparin for > 2 weeks at the time of randomization; subjects on therapeutic or prophylactic anticoagulation including warfarin will have PTT and INR as determined by the Investigator; prophylactic use of an anticoagulant to maintain patency of a vascular access device is also allowed)
* Serum creatinine =< 2.0
* Creatinine clearance > 60 ml/min
* Left ventricular ejection fraction (LVEF) > lower limit of normal (LLN) on multi gated acquisition scan (MUGA)
* Ability to understand and willingness to sign a written informed consent document
* Ability to take oral medication
* Fasting serum cholesterol < 300 mg/dL and triglycerides < 2.5 x ULN; Note: in case one or both of these thresholds are exceeded, the patient can be included after initiation of appropriate lipid lowering medication if on repeat analysis, both levels fall within parameters
* Able and willing to comply with testing and treatment as outlined in this protocol

Exclusion Criteria:

* Patients with more than one prior chemotherapy regimen for management of primary disease
* Patients who have received a prior mammalian target of rapamycin (mTOR) inhibitor
* Chronic treatment with systemic steroids or other immunosuppressive agents; Note: topical or inhaled steroids are allowed
* Uncontrolled brain or leptomeningeal metastases, including those who continue to require glucocorticoids for brain or leptomeningeal metastases
* Other malignancies =< 3 years prior to registration except for adequately treated carcinoma of the cervix or basal or squamous carcinomas of the skin
* Other concurrent severe and/or uncontrolled medical disease which could compromise participation in the study; examples include, but are not limited to: uncontrolled diabetes defined as fasting serum glucose > 1.5 x ULN; uncontrolled hypertension, or greater than 150/100 in spite of antihypertensive therapy; active (acute or chronic) or uncontrolled severe infection; unstable angina pectoris, symptomatic congestive heart failure (New York Heart Association Class III or IV); ventricular arrhythmias, active ischemic heart disease, myocardial infarction within six months; liver disease such as cirrhosis, chronic active hepatitis or chronic persistent hepatitis
* Known history of human immunodeficiency virus (HIV) seropositivity as these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy and the potential pharmacokinetic interaction between antiretroviral therapy and the investigational agent
* Known history of Hepatitis B or C as these patients may be at risk of disease reactivation when treated with the chemotherapy and/or the investigational agent
* Patients should not receive immunization with attenuated live vaccines =< 7 days of study entry or during study period
* Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of RAD001 (i.e. ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or small bowel resection sufficient to impair absorption of drug)
* Patients with clinical symptoms of gastrointestinal obstruction and who require parenteral hydration/nutrition
* Patients with an active bleeding diathesis
* Women who are pregnant or breast-feeding, or women able to conceive and unwilling to practice an effective method of birth control; (women of childbearing potential must have a negative urine or serum pregnancy test within =< 7 days prior to administration of RAD001); oral, implantable or injectable contraceptives may be affected by cytochrome P450 interactions and are therefore not considered effective for this study
* History of noncompliance with medical regimens
* Patients with a known hypersensitivity to any of the study agents
* Patients unwilling or unable to comply with the outlined protocol
* Patients with psychiatric illness or social situations that would limit compliance with study requirements

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2010-12-14 (Actual); Primary Completion 2018-01-08 (Actual); Study Completion 2018-01-08 (Actual)

PRIMARY OUTCOMES:
MTD of RAD001 in combination with carboplatin and pegulated liposomal doxorubicin | About 24 weeks
  Determine the MTD of RAD001 (everolimus) in combination with carboplatin and pegylated liposomal doxorubicin. The MTD is defined as the dose level closest to, but not over that which is predicted to result in a DLT rate of 30%, the target toxicity.

SECONDARY OUTCOMES:
Safety/tolerability of the three drug combination of carboplatin, PLD and RAD001 based on Common Terminology Criteria for Adverse Events (CTCAE) v4.0 | Every 28 days and when patient is removed from study for any reason
  Determine safety/tolerability of the three drug combination of carboplatin, PLD and RAD001. Determine preliminary analysis of anti-tumor activity of this regimen in patients with recurrent ovarian, fallopian tube or primary peritoneal cancers.
Preliminary analysis of anti-tumor activity of this regimen in patients with recurrent ovarian, fallopian tube or primary peritoneal cancers | Baseline and every 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Gina Martina-Smaldone, MD, Principal Investigator — Fox Chase Cancer Center
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States